CLINICAL TRIAL: NCT04769674
Title: Effectiveness Study of STAR (Sensory Therapies and Research) Intervention for School-Based Occupational Therapy Services for Students With Sensory Processing Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Colleen Cameron Whiting, Primary Investigator, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5722E
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Sensory Processing Disorder

STUDY DESIGN:
Intervention Model Description: Multiple baseline design across participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAR intervention (Experimental): Each research participant will receive individual 30-minute therapy sessions two times per week for fifteen weeks. Fifteen weekly ten-minute consultations with the teacher will also be conducted for each participant.
  Interventions: Other: Sensory Integration Intervention through the STAR Frame of Reference

INTERVENTIONS:
Other: Sensory Integration Intervention through the STAR Frame of Reference — The individualized therapy program will be based on the results of the comprehensive evaluation. Intervention aligns with the STAR Frame of Reference fidelity measure and Ayres Fidelity Measure.

SUMMARY:
The multiple baseline single subject design study with replication across three participants in a public-school setting. The 15-week independent variable will be a direct service occupational therapy intervention, combined with teacher consultations, based on the STAR (Sensory Therapies and Research) Frame of Reference. Frequently measured dependent variables, as the main determinants of change resulting from the intervention, will be student's video-recorded performance in the areas of functional regulation and active participation in the classroom, as rated by a trained observer. Findings of the single subject study will be corroborated via semi-structured interviews with the student participants and their teachers, administration of systematic assessments and Goal Attainment Scaling.

ELIGIBILITY:
Inclusion Criteria:

1. Student has a) suspected sensory processing challenges and b) difficulty with functional regulation and active participation in the classroom.
2. not remediated by Tier 2 intervention
3. Evaluation finds:

   1. total score, or 3 or more scales, for the main classroom on the Sensory Processing Measure are more than one standard deviation, namely is in the some problems or definite difference range,
   2. clinical determination that the student demonstrates disrupted sensory processing issues that are impacting his or her ability to participate in the school setting, and
   3. student requires specialized intervention in the form of direct pull-out service delivery in order to access his or her education.

Exclusion Criteria:

1. The student has an autism diagnosis or a primary genetic, orthopedic, or neurological disorder.
2. The student is participating in occupational therapy outside of school.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Repeated Dependent Variable Measurement | 5-7 weeks of Baseline and 15 weeks of intervention for a total of up to 22 weeks
  Repeated dependent variable measurement will be based on weekly video recorded samples of functional regulation and active participation behaviors in the classroom rated by a trained observer. Each student participant will be videotaped while in the general education classroom for 10 minutes once per week.

SECONDARY OUTCOMES:
Behavior Assessment System for Children-3 (BASC-3) | During first week of baseline and again within a week of completion of 15 weeks of intervention
  The Behavior Assessment System for Children -3, as a teacher rating scale, is a tool that measures the student's adaptive and problem behaviors in the school setting. Scores will not be compared but general clinical categories that can be rated as normal, at risk or clinically significant.
Short Child Occupational Profile (SCOPE) | During first week of baseline and again within a week of completion of 15 weeks of intervention
  The Short Child Occupational Profile is a 25-item word-based occupation-focused assessment that measures components based on the Model of Human Occupation (MOHO) and was designed to provide a broad overview of a child's occupational participation. Total scores will be between 0 and 57. A higher score will be better, indicating better function.
Goal Attainment Scaling (GAS) | During first week of baseline and again within a week of completion of 15 weeks of intervention
  A therapist who is using the Goal Attainment Scaling method with a student needs to both accurately predict the level of performance at the end of an identified period of time and decide upon what performance will look like in scaled intervals above and below the expected level of goal attainment. The teacher and occupational therapist then will develop the goal attainment follow-up guide in which expected level of achievement for each goal is scaled as zero, and achievement above and below is scaled from -2 to +2, to measure progress following intervention. 0 is expected performance and +2 is much more than expected.
Semi-structured interview with teacher | Within a week of completing 15 weeks of intervention
  Each participant's main classroom teachers will be interviewed in a semi-structured format to determine gains in perceived competency for supporting the students with sensory processing challenges following the last session of intervention.
Semi-structured interview with student | Within a week of completing 15 weeks of intervention
  Each student participant will have the opportunity to comment on his or her lived experience in a semi-structured interview following the last session of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Jacobs, Study Chair — Boston University
Locations (1):
- H. Olive Day School, Norfolk, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No